CLINICAL TRIAL: NCT03810820
Title: Remote ECG Monitoring to Reduce Complications Following Transcatheter Aortic Valve Implantations
Brief Title: Remote ECG Monitoring of TAVI Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Southlake Regional Health Centre (Other); Sunnybrook Health Sciences Centre (Other); M-Health Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REdireCT TAVI
Record Dates: First submitted 2018-11-02; First posted 2019-01-22 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Valve Disease; Aortic Valve Stenosis
Keywords: TAVR; TAVI; Heart block; Atrial fibrillation; Cardiac arrhythmias; Permanent pacemaker; Remote cardiac monitoring; Loop monitor
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Heart Block; Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Prospective cohort of consecutive patients booked for outpatient TAVI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outpatient TAVI (Other): Consecutive patients scheduled for outpatient TAVI.
  Interventions: Device: mobile Cardiac Arrhythmia Diagnostics Service (m-CARDS)

INTERVENTIONS:
Device: mobile Cardiac Arrhythmia Diagnostics Service (m-CARDS) — A wearable cardiac monitoring device is provided to patients pre- and post-TAVI. The monitor transmits cardiac data in real time to the m-CARDs team. Cardiac abnormalities are reported to the clinical team who then assess the abnormality and intervene as clinically necessary.

SUMMARY:
After surgery, patients who undergo transcatheter aortic valve implantation (TAVI) are at risk of developing cardiac arrhythmias such as heart blocks and atrial fibrillation. Current practice is to monitor TAVI patients in hospital for 2-8 days post procedure using scarce and expensive hospital telemetry beds. This study will use a new monitoring service called mobile Cardiac Arrhythmia Diagnostics Service (m-CARDS) to risk stratify patient pre-TAVI and provide an added layer of monitoring that would support earlier discharge of suitably identified patients 24-hours post TAVI. The study will assess whether this strategy will significantly reduce the pressure on hospital resources while improving patient outcomes and experience.

DETAILED DESCRIPTION:
Aortic stenosis (AS), the most common valvular heart disease, occurs when there is a narrowing of the aortic valve opening. New transcatheter aortic valve implantation (TAVI, also called transcatheter aortic valve replacement [TAVR]), is a minimally invasive surgical procedure that is rapidly expanding as the dominant treatment modality for elderly patients with AS. Approximately 1000 patients will undergo TAVR surgery in Ontario in fiscal year 2018-2019 and that number is expected to increase to ~80% of all valve replacement surgery within the next 5 years.

Patients that undergo TAVI are at risk of developing cardiac arrhythmias such as heart block and atrial fibrillation and many are routinely monitored in-hospital for 5-8 days post-surgery. Currently, this monitoring is done using scarce and expensive hospital telemetry beds.

This study uses a novel clinical pathway including remote monitoring pre- and post-TAVI using a new service called mobile Cardiac Arrhythmia Diagnostics Service (m-CARDS™). m-CARDS™ consists of a patient cardiac monitoring device that transmits cardiac data in real time to a centralized center. Patients wearing the device can remain in the comfort of their own home while being monitored remotely. The monitoring device is Health Canada approved and has been used extensively. Because it is highly sensitive to cardiac arrhythmias, including all levels of heart block, it is ideally suited for this type of monitoring.

If this pathway is adopted across all centres it will significantly reduce the pressure on hospital resources while at the same time improve the patient experience, enabling them to get home sooner. Hospital telemetry is very expensive. Reducing the length of stay from 2-8 days on average to 24hr for many patients would represent cost savings to the hospitals and province.

While some studies show that patients could be discharged earlier, there is still significant variability in adopting a short length of stay post-TAVI due to a perceived need for inpatient monitoring and lack of adequate knowledge and data on feasibility of remote outpatient monitoring.

In addition, the pre-TAVR monitoring will enhance our ability to predict and plan for interventions such as permanent pacemaker implantation. The primary objective of this project will be to facilitate the implementation of this monitoring technology into a busy tertiary care setting and better understand the conditions necessary for successful implementation. This will be achieved through ongoing stakeholder engagement (patient, provider, and hospital administrators) at all stages of the implementation program and close evaluation of quality metrics to ensure fidelity of the m-CARDS™ system.

Overall, implementation of this system is expected to impact the following levels of the health care system:

i) Patient-Level: Improved quality of life through "better care closer to home" facilitated by physician supported monitoring before TAVI and post-TAVI discharge from hospital.

ii) Provider-Level/Organizational-Level: Integrate the m-CARDS™ system into a busy TAVI clinical care pathway that can be adapted at other TAVI centres and ensure physician/administrator engagement/confidence in this novel technology.

iii) System-Level: Reduced (1) hospital length of stay and associated costs, (2) readmissions and unplanned medical visits, and (3) likelihood of hospital acquired infections.

ELIGIBILITY:
Inclusion Criteria:

* All patients selected for TAVI procedure that do not meet exclusion criteria and provide informed consent.

Exclusion Criteria:

* Patients with prior PPM or ICD
* Patient in-hospital awaiting TAVI
* Resting 12-lead ECG shows first degree AV block, plus LAHB plus RBBB; high grade 2nd or 3rd degree heart block

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment rate | End of study (Approximately Month 24)
  To achieve recruitment of at least 80% of eligible patients and to describe reasons for non-participation.
Feasibility: Participant adherence to monitoring pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  To achieve patient level adherence to monitoring at least 80% of the expected time (total # of days (hours) of loop monitoring pre-TAVI).
Feasibility: Participant adherence to monitoring post-TAVI | End of post-TAVI monitoring period (approximately Month 2 dependent on scheduling of TAVI procedure)
  To achieve patient level adherence to monitoring at least 80% of the expected time (total # of days (hours) of loop monitoring post-TAVI).
Feasibility: Requirement for PPM pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  Pre-TAVI identification of at least 5-10% of the cohort population who would need permanent pacemaker (either heart block or characteristics high risk for heart block).
Feasibility: Participant adherence to post-TAVI monitoring protocol | End of post-TAVI monitoring period (approximately Month 2)
  To facilitate complete success with post-discharge monitoring in > 80% of recruited and eligible participants (wearing monitor on same day as discharge for at least one week).
Feasibility: Timeliness of medical assessment of participants with "serious" arrhythmia identified on monitor pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  To have 80% rate of medical assessment within 24 hours for any recruited and eligible patients with identified "serious" arrhythmia pre-TAVI.
Feasibility: Timeliness of medical assessment of participants with "serious" arrhythmia identified on monitor post-TAVI | End of post-TAVI monitoring period (approximately Month 2)
  To have 80% rate of medical assessment within 24 hours for any recruited and eligible patients with identified "serious" arrhythmia post-TAVI.
Patient Experience Questionnaire | 30-day follow-up
  Survey of patient experience related to shortened length of hospital stay due to remote ECG monitoring via loop monitor and experience of care given when there are clinical findings on loop monitor
Clinical Team Experience Questionnaire | 30-day follow-up
  Survey of clinical team experience related to implementation of a new clinical pathway for pre- and post-procedure care of TAVI patients.
Number of participant or clinical team activations based on monitor findings pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  Total number of clinical team and participant activations, along with a) Inappropriate clinical team and participant activations - clinical team is activated but no patient intervention is undertaken and b) Inappropriate negative activations - arrhythmia event is seen on loop monitoring but clinical team is not activated.
Number of participant or clinical team activations based on monitor findings post-TAVI | End of post-TAVI monitoring period (approximately Month 2)
  Total number of clinical team and participant activations, along with a) Inappropriate clinical team and participant activations - clinical team is activated but no patient intervention is undertaken and b) Inappropriate negative activations - arrhythmia event is seen on loop monitoring but clinical team is not activated.
Time from identification of findings on remote monitor to clinical team activation for pre-TAVI findings. | End of pre-TAVI monitoring period (Day 14)
  Time from when a finding is noted on remote monitor to the time the clinical team is activated to assess and intervene with the participant.
Time from identification of findings on remote monitor to clinical team activation for post-TAVI findings. | End of post-TAVI monitoring period (approximately Month 2)
  Time from when a finding is noted on remote monitor to the time the clinical team is activated to assess and intervene with the participant.

SECONDARY OUTCOMES:
Hospital length of stay post-TAVI | Month 2 (approximate, dependent on scheduling of TAVI procedure)
  Duration of hospitalization post-TAVI procedure.
Arrhythmia-related unplanned re-hospitalization | 30-day post-TAVI follow-up assessment
  Unscheduled hospitalization or prolongation of hospitalization for heart rhythm reasons or PPM insertion pre- or post-TAVI.
New onset of advanced AVB pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  Defined as 2:1 second-degree or higher AVB.
New onset of advanced AVB post-TAVI | End of post-TAVI monitoring period (approximately Month 2)
  Defined as 2:1 second-degree or higher AVB.
New onset paroxysmal AF pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  Defined as any irregular atrial rhythm with absence of consistent P waves lasting > 6 seconds.
New onset paroxysmal AF post-TAVI | End of post-TAVI monitoring period (approximately Month 2)
  Defined as any irregular atrial rhythm with absence of consistent P waves lasting > 6 seconds.
New onset atrial tachycardia pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  Defined as period of sudden rapid and regular atrial rhythm with identifiable P waves.
New onset atrial tachycardia post-TAVI | End of post-TAVI monitoring period (approximately Month 2)
  Defined as period of sudden rapid and regular atrial rhythm with identifiable P waves.
New onset NSVT pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  Defined as runs of >/= 3 ventricular beats at a heart rate of > 100 bpm lasting < 30 seconds.
New onset NSVT post-TAVI | End of post-TAVI monitoring period (approximately Month 2)
  Defined as runs of >/= 3 ventricular beats at a heart rate of > 100 bpm lasting < 30 seconds.
New sustained VT pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  Defined as ventricular runs lasting >/= 30 seconds.
New sustained VT post-TAVI | End of post-TAVI monitoring period (approximately Month 2)
  Defined as ventricular runs lasting >/= 30 seconds.
Severe bradycardia pre-TAVI | End of pre-TAVI monitoring period (Day 14)
  Defined as heart rate < 40 bpm.
Severe bradycardia post-TAVI | End of post-TAVI monitoring period (approximately Month 2)
  Defined as heart rate < 40 bpm.
New onset persistent LBBB | Month 2 (approximate, dependent on scheduling of TAVI procedure)
  Defined as new onset LBBB after TAVI that persisted at hospital discharge.
Temporary PM required post-TAVI | Month 2 (approximate, depending on scheduling of TAVI procedure)
  Temporary PM not removed within 4 hours of completion of leaving procedure room.
Total number of PPM implantations | 30-day post-TAVI follow-up
  Total number of PPM implantations that are either planned (if the inciting heart rhythm was identified on monitor and implantation of PPM was arranged) or unplanned (if the monitor was not the initiating factor).
Total hospitalization days up to 30 days post-TAVI | 30-day post-TAVI follow-up
  Number of days in hospital after discharge from TAVI procedure.
Emergency Department (ED) Visits | 30-day post-TAVI follow-up
  Number of ED visits.
Health care utilization costs | 30-day post-TAVI follow-up
  Costs associated with length of stay, ED use, re-admission to hospital and outpatient clinic visits will be calculated.
Syncope requiring medical assessment | 30-day post-TAVI follow-up
  Any incident of syncope that requires medical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Madhu Natarajan, M.D., Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton Health Sciences Corporation - Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natarajan MK, Sheth TN, Wijeysundera HC, Chavarria J, Rodes-Cabau J, Velianou JL, Radhakrishnan S, Newman T, Smith A, Wong JA, Schwalm JD, Duong M, Mian RI, Bishop MG, Healey JS. Remote ECG monitoring to reduce complications following transcatheter aortic valve implantations: the Redirect TAVI study. Europace. 2022 Oct 13;24(9):1475-1483. doi: 10.1093/europace/euac042. PMID 35699482